CLINICAL TRIAL: NCT06695234
Title: Effects of a Second-generation Mindfulness-based Intervention on Quality of Life, Pain Management, and Psycho-spiritual Wellbeing in Cancer Patients: A Randomised Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Derby (Other)
Responsible Party: Principal Investigator, Chloe Wells, PhD Student, University of Derby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ETH2324-3460
Record Dates: First submitted 2024-11-13; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Cancer; Mindfulness-based Intervention; Meditation; Psychological Well-Being; Spiritual Wellbeing
Keywords: mindfulness-based intervention; Cancer; mental health; wellbeing; spiritual wellbeing; second-generation mindfulness-based intervention; RCT; oncology; psycho-oncology; meditation awareness training; MAT; MBI
MeSH Terms: conditions — Neoplasms; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A 2 (Group: Intervention vs. Treatment-as-usual Control) x 4 (Time Points: baseline, week 4, week 9 post-intervention and six-month follow-up) design will be adopted.
  Those in TAU group will be offered the intervention once the study is complete.
  Qualitative interviews will be conducted with randomly selected participants from MAT intervention group, at one month follow-up and 6 month follow-up.
  Those in MAT group invited to submit weekly online diary entries throughout the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAT RCT study (Experimental): MAT vs Treatment-as- usual RCT
  Interventions: Behavioral: Meditation Awareness Training
- Qualitative follow-up (No Intervention): Qualitative follow up of a sub-sample of those within the intervention group

INTERVENTIONS:
Behavioral: Meditation Awareness Training — A second-generation mindfulness-based intervention that reincorporates Buddhist wisdom concepts into mindfulness-based intervention.
  Arms: MAT RCT study

SUMMARY:
Background This study explores the effectiveness of Meditation Awareness Training (MAT), a second-generation mindfulness-based intervention, in enhancing quality of life, pain management, and psycho-spiritual wellbeing among cancer patients. Existing research underscores the benefits of mindfulness-based interventions (MBIs) in alleviating psychological distress and improving overall quality of life for cancer patients. However, first-generation MBIs often exclude traditional Buddhist concepts such as impermanence and emptiness, Consequently, this can result in a superficial application that may not fully engage with the underlying causes of psychological distress or promote long-term spiritual and psychological growth.

In contrast, second-generation MBIs like MAT aim to reintegrate these wisdom principles, potentially offering deeper psycho-spiritual benefits. By incorporating concepts like impermanence and emptiness, these interventions encourage a more holistic understanding and acceptance of life's challenges, fostering meaningful perspectives on illness and enhancing both spiritual and psychological wellbeing. This approach seeks to provide a more comprehensive and transformative experience for individuals, particularly those facing serious health challenges such as cancer.

Aims

The primary aim is to understand the effectiveness of MAT in individuals diagnosed with cancer. The study focuses on:

Evaluating the impact of MAT on reducing psychological distress and enhancing pain management and quality of life.

Exploring whether practising Buddhist wisdom concepts can foster meaningful perspectives on illness and life, thereby increasing spiritual wellbeing.

Determining if MAT participation leads to the establishment of new daily practices and habits among cancer patients.

Method

The study employs a mixed-methods approach across three phases:

Phase 1: A quantitative study using a randomised controlled trial (RCT) design. Participants will be divided into an intervention group (MAT) and a treatment-as-usual (TAU) control group. The effectiveness of MAT will be assessed using psychometric scales at multiple time points (baseline, week 4, week 9 post-intervention, and six-month follow-up). Importantly, participants in the TAU group will be offered the MAT intervention after the completion of the RCT, ensuring that all participants have access to the potential benefits of the intervention.

Phase 2: A qualitative exploration using Interpretative Phenomenological Analysis (IPA) to gain insights into participants' lived experiences post-MAT intervention. This phase involves semi-structured interviews conducted at one month and six months post-intervention.

Phase 3: A content analysis of diary entries collected from participants during the intervention to capture real-time reflections and experiences.

Expected Outputs The study aims to provide empirical evidence on the effectiveness of MAT in improving psychological and spiritual wellbeing among cancer patients. It is expected to offer insights into how Buddhist wisdom can be integrated back into clinical mindfulness practices to enhance their impact. The findings could inform clinical practices and contribute to the development of more holistic mindfulness-based interventions for cancer care.

Project Timelines Recruitment: Began in November 2024. Phase 1: The RCT is aimed to begin in the first quarter of 2025, with the intervention lasting 8 weeks, followed by data collection at specified time points.

Phase 2: Conduct interviews at one month and six months post-intervention. Phase 3: Collect and analyse diary entries throughout the 8-week intervention. The entire study is structured to ensure comprehensive data collection and analysis, allowing for both quantitative and qualitative insights into the MAT intervention's impact on cancer patients.

DETAILED DESCRIPTION:
Spiritual wellbeing has been shown to contribute to quality of life in cancer patients, with the National Institute for Health and Care Excellence (NICE) implementing spiritual wellbeing support as part of their person-centred care initiative (NICE, 2004). A cancer scare and diagnosis can lead to individuals contemplating their mortality and life perspective, regardless of whether they receive a palliative prognosis, they are invariably reminded of human vulnerabilities to disease, death and suffering. During contemplation, many patients begin questioning what their life is about and whether they have spent their time 'wisely' (Vehling & Phillipp, 2018).

Mindfulness is a meditative technique that derives from Buddhist practice and refers to an individual remaining 'present' attentionally, with the notion that they can embrace life as it is in that moment (Sapthiang et al., 2023). The effectiveness of mindfulness-based interventions (MBIs) in enhancing the wellbeing of individuals diagnosed with cancer, particularly in reducing anxiety and depression levels, and improving overall quality of life, has been documented in studies (Chayadi et al., 2020; Shennan et al., 2011). Moreover, research conducted by the current PhD candidate (Wells et al., 2020) has further confirmed these benefits by demonstrating significant reductions in anxiety and depression scores among cancer patients who underwent an 8-week Mindfulness-Based Cognitive Therapy (MBCT) intervention. However, the rapidness with which MBIs have been adopted and rolled out amongst clinical settings and populations have raised concerns as to whether these interventions encompass the 'true' meaning of the concept of mindfulness. For example, researchers have suggested that First-Generation MBIs (FG-MBIs), such as Mindfulness-Based Cognitive Therapy (MBCT) and Mindfulness-Based Stress Reduction (MBSR), have been tailored towards Western perspectives and thus overlook important Buddhist wisdom concepts. Examples of such wisdom principles include emptiness and impermanence, which have been shown to enhance effective mindful practice and increase personal spirituality (Shonin et al., 2014).

This critique of FG-MBIs led to the investigation of second-generation MBIs (SG-MBIs), including Meditation Awareness Training (MAT). MAT is based on the idea that mindfulness is a psychospiritual intervention rather than a purely psychological one, in contrast to most FG-MBIs (Van Gordon et al., 2015). MAT includes meditative teachings and practices based on Buddhist wisdom principles such as emptiness, impermanence, and non-duality, which can cultivate deeper insights into reality and the self (Van Gordon, 2017). Empirical studies have demonstrated the efficacy of MAT in treating clinical populations, including those with pain disorders, schizophrenia, depression, anxiety, stress disorders, and addictions (Van Gordon, 2017). However, while SG-MBIs like MAT show promise for mindfulness research, findings related to clinical applications are still at an early stage, particularly for those diagnosed with cancer. Individuals with cancer often confront questions about their mortality and future suffering, leading to existential-related concerns (Puchalski, 2012). Although SG-MBIs may not provide immediate answers to these concerns, they could guide individuals to reframe negative experiences/thoughts by learning spiritual concepts such as emptiness, non-duality, and impermanence. MAT's focus on spiritual well-being makes it a promising candidate for those with cancer experiencing psychological distress and existential contemplative thoughts.

Participants in the study will be randomly assigned to one of two groups:

Intervention Group: Participants in this group will receive Meditation Awareness Training (MAT).

Control Group: Participants in this group will continue with their usual treatment without any additional intervention. Importantly, once the RCT is complete, participants in the control group will be offered the opportunity to receive MAT, ensuring everyone has access to the potential benefits of the intervention.

Participants will be assessed at four different time points:

Baseline: Before the intervention begins. Week 4: Midway through the intervention. Week 9: At the end of the intervention. Six-month Follow-up: To see if the effects last over time. What We Are Measuring

The researchers are interested in several aspects of well-being, including:

Psychological Well-being: How participants feel emotionally and mentally. Pain Severity: How much pain participants are experiencing. Quality of Life: Overall satisfaction with life and daily functioning. Spiritual Well-being: Sense of peace and purpose. Trait Mindfulness: The ability to be present and aware in the moment.

To measure these, the study will use four questionnaires:

Five Facet Mindfulness Questionnaire: Assesses mindfulness traits. FACIT-Sp: Measures spiritual well-being. McGill Pain Questionnaire Short-form: Evaluates pain levels. DASS (Depression Anxiety Stress Scales): Assesses emotional states like depression, anxiety, and stress.Additionally, researchers will look at whether changes in depression, anxiety, and stress are not only statistically significant but also meaningful in a real-world, clinical sense.

Beyond the numbers, researchers will also gather qualitative data to capture participants' personal experiences and perspectives. This might include interviews or open-ended survey questions, providing a richer understanding of how MAT affects their lives.

Researchers will also collect demographic information such as age, sex, ethnicity, educational background, and details about cancer type and stage.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over the age of 18 and have received a cancer diagnosis, including any recurrences, within the last 24 months. Eligible diagnoses can range up to, but not exceed, stage 3 cancer at the start of the study.
* Participants to be available to attend weekly 2-hour sessions for 8 weeks
* Due to the nature of the online course, participants must have access to the Internet and use an electronic device capable of joining a video conference.

Exclusion Criteria:

* Those with a palliative diagnosis
* Those who may not speak English fluently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety, Stress scale (DASS) | From enrolment, throughout the 8-week RCT, at 9 week follow up and at 6 months follow up
  Assesses emotional states like depression, anxiety, and stress. 4-point likert scale with 0 'Does not apply to me at all' to 3 ' Applies all the time'. Higher total scores indicate higher levels of each sub category, anxiety, depression and stress.
McGill Pain Questionnaire Short-form | From enrolment, throughout the 8-week RCT, at 9 week follow up and at 6 months follow up
  Evaluates pain levels. Rates 15 pain descriptors on a scale of 0-3, where 0 = none, 1 = mild, 2 = moderate, and 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the descriptors
The Functional Assessment of Chronic Illness Therapy - Spiritual Well-being Scale (FACIT-Sp) | From enrolment, throughout the 8-week RCT, at 9 week follow up and at 6 months follow up
  To measure spiritual wellbeing and overall quality of life.scored on a 5-point Likert scale, with 0 representing "not at all" and 4 representing "very much". Possible scores range from 0 to 48, with higher scores reflecting greater spiritual well-being and QOL.

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire (FFMQ) | From enrolment, throughout the 8-week RCT, at 9 week follow up and at 6 months follow up
  Used to measure mindfulness. The 39 items of the FFMQ are rated on a 5-point Likert scale, ranging from 1 (never or very rarely true) to 5 (very often or always true).igher scores indicate greater mindfulness

CONTACTS AND LOCATIONS:
Locations (1):
- University of Derby, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
In my study, I have indicated a plan to share individual participant data (IPD) because I am committed to promoting transparency and reproducibility in research. By making anonymized IPD and related data dictionaries available to other researchers after the study's completion
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Up to seven years post publication
Access Criteria: Access to the data will be granted upon request to researchers who provide a detailed proposal outlining the intended use of the data. An ethics committee will review proposals to ensure they align with ethical standards, particularly regarding participant confidentiality and the intended use of the data for advancing research in mindfulness-based intervention

REFERENCES:
- [Background] Shonin E, Van Gordon W, Griffiths MD. Meditation awareness training (MAT) for improved psychological well-being: a qualitative examination of participant experiences. J Relig Health. 2014 Jun;53(3):849-63. doi: 10.1007/s10943-013-9679-0. PMID 23377964
- [Background] Van Gordon W, Shonin E, Griffiths MD. Towards a second generation of mindfulness-based interventions. Aust N Z J Psychiatry. 2015 Jul;49(7):591-2. doi: 10.1177/0004867415577437. Epub 2015 Mar 23. No abstract available. PMID 25801660
- [Background] Van Gordon W, Shonin E, Dunn TJ, Garcia-Campayo J, Griffiths MD. Meditation awareness training for the treatment of fibromyalgia syndrome: A randomized controlled trial. Br J Health Psychol. 2017 Feb;22(1):186-206. doi: 10.1111/bjhp.12224. Epub 2016 Nov 25. PMID 27885763
- [Background] Van Gordon W, Shonin E, Dunn TJ, Garcia-Campayo J, Demarzo MMP, Griffiths MD. Meditation awareness training for the treatment of workaholism: A controlled trial. J Behav Addict. 2017 Jun 1;6(2):212-220. doi: 10.1556/2006.6.2017.021. Epub 2017 Apr 20. PMID 28425778
- [Background] Wells C, Malins S, Clarke S, Skorodzien I, Biswas S, Sweeney T, Moghaddam N, Levene J. Using smart-messaging to enhance mindfulness-based cognitive therapy for cancer patients: A mixed methods proof of concept evaluation. Psychooncology. 2020 Jan;29(1):212-219. doi: 10.1002/pon.5256. Epub 2019 Nov 25. PMID 31654533
- [Background] Shennan C, Payne S, Fenlon D. What is the evidence for the use of mindfulness-based interventions in cancer care? A review. Psychooncology. 2011 Jul;20(7):681-97. doi: 10.1002/pon.1819. Epub 2010 Aug 4. PMID 20690112
- [Background] Puchalski CM. Spirituality in the cancer trajectory. Ann Oncol. 2012 Apr;23 Suppl 3:49-55. doi: 10.1093/annonc/mds088. PMID 22628416
- [Background] Chayadi E, Baes N, Kiropoulos L. The effects of mindfulness-based interventions on symptoms of depression, anxiety, and cancer-related fatigue in oncology patients: A systematic review and meta-analysis. PLoS One. 2022 Jul 14;17(7):e0269519. doi: 10.1371/journal.pone.0269519. eCollection 2022. PMID 35834503

DOCUMENTS (1):
  • Informed Consent Form (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT06695234/ICF_000.pdf